CLINICAL TRIAL: NCT03531983
Title: Results of Gamma Nail in Trochentric Fractures of the Adults
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Gamal Helmy, Assistant Lecturer, Assiut University
Other Study IDs: G.nail in trochentric frs
Record Dates: First submitted 2018-04-20; First posted 2018-05-22 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Trochanteric Fractures
Keywords: gamma nail
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: fixation of tochentric fractures by gamma nail — • Thirty patients with recent traumatic extracapsular proximal femoral fractures were treated using a short gamma nail of third-generation assembly

SUMMARY:
We prospectively reviewed the results of 30 patients who had undergone intramedullary fixation with a gamma nail for femur trochentric fractures in AUH. within 1 year

DETAILED DESCRIPTION:
Hip fractures are considered one of the major health problems in aging societies . These fractures are correlated with increased disability and mortality and a decreased quality of life . Early mobilization of patients with these fractures is essential to improve fracture healing, minimize immediate postsurgical morbidity, and reduce care costs. One essential prerequisite for early mobilization is mechanically stable fracture fixation . Nowadays, most hip fractures are treated by extramedullary or intramedullary implants, which allow a stable fixation in the majority of cases

A dynamic hip screw (DHS) is the most commonly used implant for intertrochanteric fractures . Load bearing in the proximal femur is predominantly through the intact calcar femoral; the lever arm of the laterally placed plate is increased, thus, there is a risk of implant cutout if the calcar is not intact .

Biomechanically, compared with a laterally fixed side plate, an intramedullary device decreases the bending force of the hip joint on the implant by 25-30%. This has advantages especially in elderly patients, in whom the primary treatment goal is immediate full weight-bearing mobilization.

It has been postulated that cephalomedullary nails have an advantage over DHS fixation because of the load-bearing axis being closer to the hip joint fulcrum, and also less blood loss, minimal tissue dissection, shorter operation time, and faster ambulation after surgery . However, other studies have reported that fixation with DHS is better . One of the major drawbacks discovered with the use of the gamma nail is a higher reoperation rate as a result of new fracture around the implant . In this study, we present our results for the treatment of trochentric fractures using a gamma nail in terms of the outcome, drawbacks, and possible complications.

ELIGIBILITY:
Inclusion Criteria:

* Age (20-70)
* unstable trochentric fractures

Exclusion Criteria:

* pathological fractures due to neoplasia

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients who were admitted to AUH with trochentic fracture and treated by gamma nail
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with failure of initial intervention | 1 year
  case series prospective study for 30 patients who were admitted to AUH during 18-month period from December 2018 to May 2019